CLINICAL TRIAL: NCT00616161
Title: A Phase II Study to Assess the Hemodynamic Effects of Istaroxime, a Novel Lusinotropic Agent, in Patients Hospitalized With Worsening Heart Failure and a Reduced Left Ventricular Systolic Function
Brief Title: A Phase II Trial to Assess Hemodynamic Effects of Istaroxime in Pts With Worsening HF and Reduced LV Systolic Function
Acronym: HORIZON-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Collaborators: MDS Pharma Services (Industry)
Responsible Party: Mihai Gheorghiade, MD, FACC Professor of Medicine and Surgery, Associate Chief, Division of Cardiology, Northwestern University, Feinberg School of Medicine - 201 E. Huron - Chicago IL
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PST2744-DM-04-012
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Heart Failure
Keywords: Acute Heart Failure; Inotropes; Lusitropic agents; Istaroxime; PST2744
MeSH Terms: conditions — Heart Failure | interventions — Istaroxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Istaroxime dose of 0.5 microgram/kg body weight/minute of iv infusion for six ours
  Interventions: Drug: Istaroxime
- 2 (Experimental): Istaroxime dose of 1.0 microgram/kg body weight/minute of iv infusion for six ours
  Interventions: Drug: Istaroxime
- 3 (Experimental): Istaroxime dose of 1.5 microgram/kg body weight/minute of iv infusion for six ours
  Interventions: Drug: Istaroxime
- 4 (Placebo Comparator): Placebo iv infusion for six ours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Istaroxime — 0.5 microgram/kg/min IV for 6 hours
  Other Names: PST2744
  Arms: 1
Drug: Istaroxime — 1.0 microgram/kg/min IV for 6 hours
  Other Names: PST2744
  Arms: 2
Drug: Istaroxime — 1.5 microgram/kg/min IV for 6 hours
  Other Names: PST2744
  Arms: 3
Drug: Placebo — Placebo
  Other Names: placebo of PST2744
  Arms: 4

SUMMARY:
The purpose of this study is to determine the minimum effective dose of Istaroxime, in patients requiring hospitalization for deterioration of chronic heart failure and left ventricular systolic dysfunction. This goal will be reached by comparing the hemodynamic effect of three different doses of the drug versus placebo. Efficacy will be measured as a change in Pulmonary Capillary Wedge Pressure from pre-infusion to the last assessment at six hours intravenous infusion.Secondary objectives will be to evaluate safety, tolerability and efficacy on other main hemodynamic parameters, echocardiographic and echo-doppler measurements, plus preliminary pharmacokinetics of the drug.

DETAILED DESCRIPTION:
Congestive heart failure is one of the most common cardiovascular conditions and it is presently reaching epidemic proportions. The prevalence of chronic heart failure has risen specifically as a result of the increased longevity and longer survival after myocardial infarction. In 2003, over one million hospitalization with a primary diagnosis of heart failure occurred in the United States of America, and a similar number has been reported in Europe, too. At present, approximately 5 million Americans are estimated to suffer of this syndrome and the number is expected to continue to increase with the increase and aging of the population. Despite advances in treatment, the mortality remains high in U.S.A. as in Europe, with nearly three hundred thousands patients dying of CHF as the primary or contributory cause each year.

The total number of hospital admissions approaches 3 million yearly when HF is listed as a primary or secondary diagnosis. Although these patients have a relatively low mortality during the hospitalization (less than 4%), the readmission rates within 60 days of discharge range from 20 to 30% and mortality within 60 days of discharge is 5 - 10%.

The primary aim of acute treatment of worsening CHF is to alleviate the symptoms of congestion and edema, improve the hemodynamic profile, and preserve renal function without causing myocardial injury. Improved hemodynamics usually results in relief of primary symptoms like dyspnea and edema and in a consequent improved sense of wellbeing and mental status. The improvement in hemodynamics may persist after the pharmacological interventions used in the acute phase are withdrawn.

The need in this setting is to decrease the filling pressures (RA pressure and PCWP), increase cardiac output, without increasing the heart rate and inducing/worsening atrial or ventricular arrhythmias. In addition, the agent should improve diastolic function, modulate the exaggerated neurohormonal responses to CHF and preserve/protect the viable but non contractile myocardium (e.g.: the hibernated myocardium). The agent should also facilitate the earlier start of life-saving therapies (e.g. beta - blockers).Pre-clinical data on Istaroxime show that this drug increases contractility without increasing heart rate and oxygen consumption; furthermore it is improving diastolic dysfunction and it not causing vasodilatation.

ELIGIBILITY:
Inclusion Criteria:

* Signing of a written informed consent form.
* Male or female patients aged between 18 and 85 years.
* Negative pregnancy test at screening, for women of childbearing potential.
* Body weight less or equal to 100 kg.
* Blood pressure not more than SAP=150 or DAP=90 mmHg.
* Heart rate in the range of 60-110 bpm
* Adequate Echo window available.
* Hospital admission to a monitored bed with a primary diagnosis of worsening of heart failure and LV Ejection Fraction less or equal to 35% documented by 2D-Echocardiogram, or radionuclide angiography or LV angiogram within 6 months prior to screening or at hospitalization.
* the clinical condition of the patient are stabilized within 48 hours from hospitalization and do not require continuous iv drug treatments
* no need for additional new oral treatments or any intravenous treatment administration over the following 8 hours is foreseen

Randomisation period inclusion criteria:

* Any residual sign of heart failure (e.g.: Jugular Venous Distension, and/or Rales and/or Peripheral Oedema) associated with a PCWP more or equal to 20 mmHg,
* The last three consecutive determinations of PCWP, obtained during the stabilization period, have to be in a maximum range of variability of 10%.

Exclusion Criteria:

* Ongoing treatment with oral or intravenous inotropes and/or inodilators.
* Patient treated with digoxin within the last week, can be randomised if the plasma concentration of digoxin are tested before randomisation and its value will be less than 0.5 ng/ml.
* Intermittent inotropes administration within 2 weeks.
* Symptoms of Heart Failure at randomization e.g.: dyspnoea
* Systolic blood pressure < 90 mmHg.
* Atrial fibrillation within 2 weeks.
* Left Ventricular Bundle Branch Block
* Cardiogenic shock or mechanical ventilation.
* Creatinine level > 3.0 mg/dl or requiring dialysis treatment.
* Left ventricular failure primarily from uncorrected obstructive valvular disease, hypertrophic obstructive cardiomyopathy, restrictive/obstructive cardiomyopathy, uncorrected thyroid disease, known acute myocarditis, known amyloid cardiomyopathy.
* Artificial heart valve.
* Electrical device implanted (ICD, CRT)
* Evidence of acute coronary syndrome within 3 months.
* History of stroke or transient ischemic attack in the 6 months prior to screening.
* History of sustained ventricular tachycardia.
* Coronary by-pass grafting or PTCA within the last 30 days
* INR > 1.5.
* Status post successful cardiac resuscitation.
* Serum K < 3.5 mEq/l or > 5.3 mEq/l just prior to treatment.
* ALT, AST > 3 times the upper normal limit just prior to treatment.
* Hemoglobin < 10 g/dl (either gender) just prior to treatment.
* Other clinically significant laboratory or medical conditions, which in the opinion of the Investigator make the patient unsuitable for evaluation in the study.
* Anticipated survival of less than 2 months for concomitant diseases.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To determine the minimum effective dose of ISTAROXIME by comparing the hemodynamic effect of 3 different doses of the drug versus placebo. Efficacy will be measured as a change in PCWP from right heart catheterization. | 6 hours drug infusion

SECONDARY OUTCOMES:
safety, tolerability and efficacy on blood pressure, heart rate, cardiac index, stroke work index, right atrial pressure, systemic and pulmonary vascular resistances, Echocardiographic and Doppler parameters, neurohormonal parameters and renal function. | 6 and 24 hours after start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Gheorghiade, MD FACC, Study Chair — Northwestern University Feinberg School of Medicine - Chicago; Witold Ruzyllo, MD, Principal Investigator — National Institute of Cardiology, Department of Coronary Artery Disease - Warsaw - POLAND; Cezar Macarie, MD, Principal Investigator — Insitutul de Boli Cardiovasculare C.C. Iliescu Bucuresti, Bucharest - ROMANIA; Dimitrios Th Kremastinos, MD, Principal Investigator — Second Cardiology Department, Athens University Medical School, University Hospital Attikon, Athens - GREECE; Serban I Bubenek-Turconi, MD, Principal Investigator — First Anaesth. & Intensive Care Dept., CC Iliescu Heart Disease Institute, Bucharest - ROMANIA; Maria Dorobantu, MD, Principal Investigator — Emergency Hospital "Loreasca", Bucharest - ROMANIA; Jerzy Korewicki, MD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Jaroslaw Drodz, MD, Principal Investigator — Hospital bieganskieko , Dept of Cardiology, Lodz - POLAND; Piotr Ponikowski, MD, Principal Investigator — Iv Military Hospital, Wroclaw, POLAND; John N Nanas, MD PhD, Principal Investigator — Alexandra University Hospital, Athens - GREECE

REFERENCES:
- [Background] Gheorghiade M, Sabbah HN. Istaroxime: an investigational luso-inotropic agent for acute heart failure syndromes. Am J Cardiol. 2007 Jan 22;99(2A):1A-3A. doi: 10.1016/j.amjcard.2006.09.001. Epub 2006 Sep 18. No abstract available. PMID 17239700
- [Background] Micheletti R, Palazzo F, Barassi P, Giacalone G, Ferrandi M, Schiavone A, Moro B, Parodi O, Ferrari P, Bianchi G. Istaroxime, a stimulator of sarcoplasmic reticulum calcium adenosine triphosphatase isoform 2a activity, as a novel therapeutic approach to heart failure. Am J Cardiol. 2007 Jan 22;99(2A):24A-32A. doi: 10.1016/j.amjcard.2006.09.003. Epub 2006 Sep 25. PMID 17239701
- [Background] Mattera GG, Lo Giudice P, Loi FM, Vanoli E, Gagnol JP, Borsini F, Carminati P. Istaroxime: a new luso-inotropic agent for heart failure. Am J Cardiol. 2007 Jan 22;99(2A):33A-40A. doi: 10.1016/j.amjcard.2006.09.004. Epub 2006 Sep 18. PMID 17239702
- [Background] Sabbah HN, Imai M, Cowart D, Amato A, Carminati P, Gheorghiade M. Hemodynamic properties of a new-generation positive luso-inotropic agent for the acute treatment of advanced heart failure. Am J Cardiol. 2007 Jan 22;99(2A):41A-46A. doi: 10.1016/j.amjcard.2006.09.005. Epub 2006 Sep 18. PMID 17239704
- [Background] Ghali JK, Smith WB, Torre-Amione G, Haynos W, Rayburn BK, Amato A, Zhang D, Cowart D, Valentini G, Carminati P, Gheorghiade M. A phase 1-2 dose-escalating study evaluating the safety and tolerability of istaroxime and specific effects on electrocardiographic and hemodynamic parameters in patients with chronic heart failure with reduced systolic function. Am J Cardiol. 2007 Jan 22;99(2A):47A-56A. doi: 10.1016/j.amjcard.2006.09.006. Epub 2006 Sep 20. PMID 17239705
- [Background] Wehrens XH. Istaroxime, a novel luso-inotropic agent for the treatment of acute heart failure. Curr Opin Investig Drugs. 2007 Sep;8(9):769-77. PMID 17729189
- [Background] Adamson PB, Vanoli E, Mattera GG, Germany R, Gagnol JP, Carminati P, Schwartz PJ. Hemodynamic effects of a new inotropic compound, PST-2744, in dogs with chronic ischemic heart failure. J Cardiovasc Pharmacol. 2003 Aug;42(2):169-73. doi: 10.1097/00005344-200308000-00003. PMID 12883318
- [Background] Ferrari P, Micheletti R, Valentini G, Bianchi G. Targeting SERCA2a as an innovative approach to the therapy of congestive heart failure. Med Hypotheses. 2007;68(5):1120-5. doi: 10.1016/j.mehy.2006.08.045. Epub 2006 Nov 17. PMID 17113239
- [Derived] Shah SJ, Blair JE, Filippatos GS, Macarie C, Ruzyllo W, Korewicki J, Bubenek-Turconi SI, Ceracchi M, Bianchetti M, Carminati P, Kremastinos D, Grzybowski J, Valentini G, Sabbah HN, Gheorghiade M; HORIZON-HF Investigators. Effects of istaroxime on diastolic stiffness in acute heart failure syndromes: results from the Hemodynamic, Echocardiographic, and Neurohormonal Effects of Istaroxime, a Novel Intravenous Inotropic and Lusitropic Agent: a Randomized Controlled Trial in Patients Hospitalized with Heart Failure (HORIZON-HF) trial. Am Heart J. 2009 Jun;157(6):1035-41. doi: 10.1016/j.ahj.2009.03.007. Epub 2009 Apr 23. PMID 19464414
- [Derived] Gheorghiade M, Blair JE, Filippatos GS, Macarie C, Ruzyllo W, Korewicki J, Bubenek-Turconi SI, Ceracchi M, Bianchetti M, Carminati P, Kremastinos D, Valentini G, Sabbah HN; HORIZON-HF Investigators. Hemodynamic, echocardiographic, and neurohormonal effects of istaroxime, a novel intravenous inotropic and lusitropic agent: a randomized controlled trial in patients hospitalized with heart failure. J Am Coll Cardiol. 2008 Jun 10;51(23):2276-85. doi: 10.1016/j.jacc.2008.03.015. Epub 2008 Apr 9. PMID 18534276